CLINICAL TRIAL: NCT00517517
Title: An Open-Label Phase I/II Study to Assess the Safety and Immunogenicity of Two Doses of a Vero Cell Derived, Whole Virus Clade 2 H5N1 Influenza Vaccine in Healthy Volunteers Aged 21 to 45 Years
Brief Title: Safety and Immunogenicity Study of Two Doses of an Inactivated H5N1 Influenza Vaccine (Whole Virion, Vero Cell Derived)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 810701
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2011-09

CONDITIONS: Influenza
Keywords: Pandemic influenza
MeSH Terms: conditions — Influenza, Human | interventions — Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intramuscular injection of whole virion, Vero cell-derived influenza vaccine containing 7.5 µg of H5N1 HA antigen per 0.5 mL in a non-adjuvanted formulation
  Interventions: Biological: Whole virion, Vero cell-derived influenza vaccine containing either 3.75 µg or 7.5 µg H5N1 hemagglutinin (HA) antigen in a non-adjuvanted formulation
- 2 (Experimental): Intramuscular injection of whole virion, Vero cell-derived influenza vaccine containing 3.75 µg of H5N1 HA antigen per 0.25 mL in a non-adjuvanted formulation
  Interventions: Biological: Whole virion, Vero cell-derived influenza vaccine containing either 3.75 µg or 7.5 µg H5N1 hemagglutinin (HA) antigen in a non-adjuvanted formulation

INTERVENTIONS:
Biological: Whole virion, Vero cell-derived influenza vaccine containing either 3.75 µg or 7.5 µg H5N1 hemagglutinin (HA) antigen in a non-adjuvanted formulation — Subjects will be randomized 1:1 to receive two intramuscular injections of the whole virion, Vero cell-derived influenza vaccine containing either 3.75 mg or 7.5 mg H5N1 hemagglutinin (HA) antigen in a non-adjuvanted formulation on Day 0 and Day 21.

SUMMARY:
The objectives of this Phase I/II study are to assess the safety and immunogenicity of two different dose levels of a non-adjuvanted H5N1 influenza vaccine in a healthy young adult population. Subjects will be randomized 1:1 to receive two intramuscular injections (21 days apart) of the vaccine containing either 3.75 µg or 7.5 µg H5N1 hemagglutinin (HA) antigen in a non-adjuvanted formulation. Subjects will be monitored for safety and for antibody response to the vaccine. A data safety monitoring board will review the safety data after the first and second vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Are 21 to 45 years of age, inclusive, on the day of screening
* Have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry
* Are clinically healthy, as determined by the Investigator's clinical judgment through collection of medical history and performance of a physical examination
* Are physically and mentally capable of participating in the study
* Agree to keep a daily record of symptoms for the duration of the study
* If female and capable of bearing children, have a negative urine pregnancy test result within 24 hours of the scheduled first vaccination and agree to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

* Have a history of exposure to H5N1 virus or a history of vaccination with an H5N1 influenza virus
* Are at high risk of contracting H5N1 influenza infection (e.g. poultry workers)
* Suffer from or have a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder
* Suffer from any inherited or acquired immunodeficiency
* Test positive for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HbsAg) or Hepatitis C Virus (HCV)
* Suffer from a disease or are undergoing a form of treatment that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs
* Have a history of inflammatory or degenerative neurological disease (e.g. Guillain Barré syndrome)
* Have a history of severe allergic reactions or anaphylaxis
* Have a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating
* Have received a blood transfusion or immunoglobulins within 90 days of study entry
* Have donated blood or plasma within 30 days of study entry
* Have received any live vaccine within 4 weeks or inactivated vaccine within 2 weeks prior to vaccination in this study
* Have undergone systemic corticoid therapy within 30 days prior to study entry
* Have a functional or surgical asplenia
* Have a known or suspected problem with alcohol or drug abuse
* Were administered an investigational drug within six weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product
* Are a member of the team conducting this study or are in a dependent relationship with the study Investigator. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site conducting the study
* If female: are pregnant or lactating

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2007-07; Primary Completion 2007-09 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with antibody response to the vaccine strain associated with protection 21 days after the second vaccination defined as titer measured by Microneutralization (MN) test >= 1:20 | 21 days after the second vaccination (= Day 42 in the study)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter Bio Science Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (4):
- Hong Kong (2):
  - University of Hong Kong, Queen Mary Hospital, Hong Kong
  - Chinese University of Hong Kong, Prince of Wales Hospital, Shatin
- Singapore (2):
  - National University Hospital, Singapore
  - Changi General Hospital, Singapore